CLINICAL TRIAL: NCT06040593
Title: Identify Predictors of Clinical Outcomes in Real-world Patients With HR+ and HER2-low/Negative Breast Cancer Treated With Neoadjuvant Chemotherapy or Endocrine Therapy
Brief Title: Study of Predictors of Clinical Outcomes in Patients With HR+ and HER2-low/Negative Breast Cancer
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: U31402-0005-NIS-EPI
Record Dates: First submitted 2023-08-28; First posted 2023-09-15 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Hormone-receptor-positive Breast Cancer; HER2-low Breast Cancer; HER2-negative Breast Cancer
Keywords: Hormone-receptor-positive Breast Cancer; HER2-low Breast Cancer; HER2-negative Breast Cancer; Real-world Data

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HR+/HER2-low Breast Cancer: Participants with HR+/HER2-low breast cancer who were treated with neoadjuvant chemotherapy or endocrine therapy identified from the ConcertAI databases.
  Interventions: Other: No drug
- HR+/HER2-negative Breast Cancer: Participants with HR+/HER2-negative breast cancer who were treated with neoadjuvant chemotherapy or endocrine therapy identified from the ConcertAI databases.
  Interventions: Other: No drug

INTERVENTIONS:
Other: No drug — This is a non-interventional study and no study drug will be provided.

SUMMARY:
There is a lack of data on clinical and patient factors that are associated with poor survival in patients with HR+ and HER2-low/negative breast cancer treated with neoadjuvant chemotherapy or endocrine therapy. This retrospective, non-interventional study is designed to assess the predictors of clinical outcomes in this patient population. No study drug will be provided as part of this study protocol.

DETAILED DESCRIPTION:
This retrospective, non-interventional study is designed to assess the following primary objectives:

1. To identify predictors of event-free survival (EFS) in patients with HR+ and HER2-low/negative breast cancer treated with neoadjuvant chemotherapy or endocrine therapy, and
2. To stratify patients according to event-free survival using different combinations of significant predictors and evaluate the patient characteristics and clinical outcomes such as EFS, overall survival and pathological complete response across patient groups of different risk level.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed HR+ and HER2-low/negative breast cancer diagnosed between January 1, 2010 and December 31, 2022 (Aged ≥18 years at the time of diagnosis)
* Stage I-IIIB at the time of diagnosis
* Received neoadjuvant chemotherapy and/or endocrine therapy and/or IO therapy
* Received curative intent surgery (mastectomy after neoadjuvant chemotherapy, endocrine, or IO therapy)

Exclusion Criteria:

* Patients who received HER2-targeted therapies including

  * Trastuzumab
  * Pertuzumab
  * Ado-trastuzumab emtansine
  * Neratinib
  * Tucatinib
  * Lapatinib
  * Fam-trastuzumab deruxtecan-nxki
  * Margetuximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HR+ and HER2-low/negative breast cancer diagnosed between January 1, 2010 and December 31, 2022 and treated with neoadjuvant chemotherapy or endocrine therapy will be identified from the ConcertAI database based on the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 927 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
Event-free survival (EFS) in Participants With HR+ and HER2-Low/Negative Breast Cancer | Index date to the end of the study period (approximately December 31, 2022)
  Events of interest include any other primary cancer, metastases, higher stage, tumor progression, and death due to any cause.
Overall Survival of Participants With HR+ and HER2-Low/Negative Breast Cancer | Index date to the end of the study period (approximately December 31, 2022)
Pathological Complete Response (pCR) in Participants With HR+ and HER2-Low/Negative Breast Cancer | Index date to the end of the study period (approximately December 31, 2022)
  Pathological complete response (pCR) was defined as ypT0/Tis ypN0 and is the absence of any invasive component in the resected breast specimen and all resected lymph nodes following completion of neoadjuvant therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- ConcertAI database, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No